CLINICAL TRIAL: NCT04171180
Title: The Efficacy of Budesonide/Formoterol in Cough Variant Asthma -- A Multi-center Randomized, Controlled Clinical Trial
Brief Title: The Efficacy of Budesonide/Formoterol in Cough Variant Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Tongji Hospital (Other); Zunyi Medical College (Other); Central South University (Other); China-Japan Friendship Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-17-13270
Record Dates: First submitted 2019-04-21; First posted 2019-11-20 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Cough Variant Asthma
MeSH Terms: conditions — Cough-Variant Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controlled group (Active Comparator): Controlled group: budesonide/formoterol(SYM) 160/4.5ug 1 inhalation bid* 3 months (n=250).
  Interventions: Drug: budesonide/formoterol
- Study group (Experimental): Study group: SYM 160/4.5ug 2 inhalation bid* 3 months (n=250).
  Interventions: Drug: budesonide/formoterol

INTERVENTIONS:
Drug: budesonide/formoterol — apply different dosage of budesonide/formoterol in two groups and evaluate the treatment effects.

SUMMARY:
Cough variant asthma (CVA), subtype of bronchial asthma, is considered to be one of the most common causes of chronic cough in different cough guidelines of United States, Europe, China and other countries. From a multicenter survey in China, over one third of chronic cough is caused by CVA, which is higher than western countries. CVA differs from classic asthma, usually manifesting a symptom of only coughing without wheezing or dyspnea and particularly coughing at night. With less clinical manifestation and medical intervention, CVA patients are easily be neglected and misdiagnosed, and 30-40% of them will develop to typical asthma in the next few years. Currently there's no specific therapy recommendation for CVA in GINA. Although cough guidelines in China recommend that CVA patients should be treated as typical asthma, no recommendation on details about ICS/LABA dosage and duration. There are only a few sporadic CVA therapy researches with small sample size. Two studiesfound that CVA patients can't get cough symptom relief even after treating by low dose of ICS/LABA for 3 months. Some patients' cough symptom relapses during the 24-week follow-up phase after treating by ICS/LABA for 3 months. Overall, the best treatment of CVA is not yet clear.

GINA 2018 emphasize that asthma need long-term management. Euro-SMART study found that budesonide/formoterol 2 inhalation twice daily plus as needed can reduce daytime asthma symptoms and night-time awakenings, as well as reduce exacerbation risk more than 1 inhalation twice daily. Based on the above reasons, We assume that increase the dosage of ICS/LABA can decrease relapse rate in CVA patients with severe cough. This multi-center, randomized, controlled clinical trial can help to clarify the best dosage of budesonide/formoterol of CVA in China.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, with age ≥18，≤70 years old.
* Diagnose with CVA
* CSS(cough symptom score, daytime + nighttime) ≥ 3 points

Exclusion Criteria:

* Participated in any interventional clinical trial during the last 90 days.
* Pregnancy
* Associated with a clear history of other lung diseases, or combined with other systems severe illness.
* A abuse history of alcohol or narcotic drug, or have a mental history, confrontation personality, adverse motives, suspicious or other emotional or intellectual problems that may affect the informed validity of the study
* With a history of upper respiratory tract infection acute exacerbation within 4 weeks before enrolment.
* Clinical abnormalities associated with symptoms in chest radiology.
* Smokers
* On medications of ACEI or ARB
* Not suitable for study observation judged by investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
the proportion of CVA patient with symptom relapse | during 6-months' follow-up phase
  Relapse rate during the 6-months' follow-up phase after treating by different doses of budesonide/formoterol for 3 months.

SECONDARY OUTCOMES:
the proportion of CVA patient with symptom relief | after treating by different doses of budesonide/formoterol for 3 months.
  symptom relief rate after treating by different doses of budesonide/formoterol for 3 months.

OTHER OUTCOMES:
change in lung function | during 6-months' follow-up phase
  value of pulmonary function index such as FEV1% Pred, FVC% Pred, PD20-FEV1 and PEF
assess different phenotypes of CVA | during 6-months' follow-up phase
  investigate inflammation characteristics consist of differential count of inflammatory cells in induced sputum
assess safety of different doses of budesonide/formoterol | during 6-months' follow-up phase
  evaluate adverse events of different doses of budesonide/formoterol

CONTACTS AND LOCATIONS:
Overall Officials: Huahao Shen, Prof., Principal Investigator — the Second Affiliated Hospital of Zhejiang University School of Medicin
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicin, Hangzhou, Zhejiang, China